CLINICAL TRIAL: NCT03821779
Title: Study of Slow Prefrontal Cortex Oscillations During Social Exposure in Social Anxiety Disorder
Brief Title: Prefrontal Oscillations in Social Anxiety Disorder (POSAD)
Acronym: POSAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C17-25
Record Dates: First submitted 2018-11-29; First posted 2019-01-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Anxiety Disorders; Anxiety; Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: First phase (go-no-go) with 10 subjects in 1 arm Second phase with 20 subjets (2 arms) in a cross-over design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Go-no-go phase (Experimental): The presence of significant prefrontal oscillations in the EEG recording 2-6Hz band during in vivo social exposure (oral presentation to examiners) will be assessed in 10 subjects with social anxiety disorder. EEG will be recorded immediately before, during and after oral presentations to examiners.
  Psychometric evaluation will be performed prior to experimental sessions. Rating of anxiety levels will be performed by subjects using a Visual Analogue Scale of anxiety during each of the 3 experimental periods (wainting, presentation, recovery).
  Results of EEG recordings in the first 10 subjects will lead to continuation (presence of significant slow prefrontal oscillations during anxiety) or interruption (absence of signification oscillation) of the study.
  Interventions: Behavioral: In vivo social exposure; Other: EEG recording; Diagnostic Test: Psychometric evaluation; Diagnostic Test: Visual Analogue Scale of anxiety
- Group 2.1 (Experimental): In group 2.1, 10 subjects will undergo 2 sessions in a cross-over design with EEG recording immediately before, during and after:
  1. "real exposure": oral presentation to a panel of examiners
  2. "virtual reality" : oral presentation to virtual examiners
  Rating of anxiety levels will be performed by subjects using a Visual Analogue Scale of anxiety during each of the 3 experimental periods for each session.
  Psychometric evaluation will be performed prior to experimental sessions.
  Interventions: Behavioral: In vivo social exposure; Behavioral: Social exposure in a virtual reality setting; Other: EEG recording; Diagnostic Test: Psychometric evaluation; Diagnostic Test: Visual Analogue Scale of anxiety
- Group 2.2 (Experimental): In group 2.2, 10 subjects will undergo 2 sessions in a cross-over design with EEG recording immediately before, during and after:
  1. "virtual reality" : oral presentation to virtual examiners
  2. "real exposure": oral presentation to a panel of examiners
  Rating of anxiety levels will be performed by subjects using a Visual Analogue Scale of anxiety during each of the 3 experimental periods for each session.
  Psychometric evaluation will be performed prior to experimental sessions.
  Interventions: Behavioral: In vivo social exposure; Behavioral: Social exposure in a virtual reality setting; Other: EEG recording; Diagnostic Test: Psychometric evaluation; Diagnostic Test: Visual Analogue Scale of anxiety

INTERVENTIONS:
Behavioral: In vivo social exposure — Subjects will be invited to give a 5 minutes oral presentation on the topic of their choice to five examiners displaying no facial emotional reaction, after a 5 minutes period of silent waiting in front of the examiners. This waiting period is prompt to elicit anticipation-type of social anxiety.
Behavioral: Social exposure in a virtual reality setting — Subjects will give a 5 minutes oral presentation on the subject of their choice to a virtual reality panel composed of 5 examiners displaying no facial emotional reaction, after a 5 minutes period of silent waiting in front of the examiners. This waiting period is expected to elicit anticipation-type of social anxiety.
  Arms: Group 2.1; Group 2.2
Other: EEG recording — EEG will be recorded with a standard 16-electrodes cap. Recordings will start before the 5 minutes waiting period and continue throughout oral presentation and recovery. The recovery period will be used as a baseline control
Diagnostic Test: Psychometric evaluation — Subjects will be evaluated prior to inclusion using the following assessment tools
  * Anamnestic Association for Methodology and Documentation in Psychiatry (AMDP) questionnaire
  * Mini International Neuropsychiatric Interview (MINI 6.0, for psychiatric diagnoses)
  * Liebowitz Social Anxiety Scale (LSAS)
  * Montgomery Asberg Depression Rating Scale (MADRS)
  * Brief Anxiety Scale of Tyrer (BAS)
  * State-Trait Anxiety Inventory (STAI A-B)
  * Global Assessment of Functioning (GAF)
Diagnostic Test: Visual Analogue Scale of anxiety — Subjects will be asked to rate their anxiety levels
  * immediately before (5 minutes of silent waiting),
  * during
  * and after the 5-minute oral presentation (recovery)

SUMMARY:
Experimental fear in rodents is correlated with slow oscillations in electrical recordings of prefrontal cortex activities. The present study aims to test whether slow prefrontal oscillations is a biomarker of pathological anxiety in human subjects.

DETAILED DESCRIPTION:
Fear and anxiety are adaptive responses that may become excessive or inappropriate in pathological conditions, as defined as anxiety disorders in DSM-5. These disorders, including phobic disorders such as social anxiety disorder, are frequent and impairing in the general population, with an estimated lifetime prevalence of 28% and significant consequences on quality of life. Direct and indirect medical costs related to these conditions amount to 74.4 billion €/year in Europe. Despite their prevalence, debilitating nature and chronicity, the pathophysiology of anxiety disorders is poorly understood and neurobiological treatments, including pharmacotherapy, are lacking efficacy. A better understanding of the neuronal mechanisms implicated in anxiety is necessary for the conception of new approaches to treat pathological anxiety.

Anxiety is commonly modeled in animals using fear conditioning, which consists in associating a neutral stimulus (eg: a sound) with a mild electrical foot-shock. As a result of the association between sound and shock, sound presentation in isolation induces a set of conditioned behavioral responses, such as an immobilization ("freezing"). Previous studies have shown that the expression of fear responses, measured on the basis of freezing, is associated with the emergence of slow oscillations (2-6Hz) in medial prefrontal cortex (mPFC) of mice. Moreover, emergence of these oscillations in mPFC is predictive of the occurrence of freezing, and the artificial induction of 4 Hz oscillations in mPFC with optogenetics induces freezing. Finally, inhibiting neurons in mPFC during the ascending phase of this slow mPFC oscillation at the time of conditioned sound presentation is sufficient to significantly reduce fear.

Interestingly, these results obtained in mice seem to find their prolongation in humans. Recent studies using fear conditioning in human subjects have also reported the emergence of prefrontal slow oscillations between 2-6 Hz during expression of conditioned fear responses. These results suggests that common mechanisms underlie the expression of fear in humans and rodents. However, whether similar neuronal circuits and mechanisms are implicated in human anxiety disorders remains unknown.

This study aims at assessing the presence of slow mPFC oscillations during expression of anxiety in patients suffering from anxiety disorders. Beyond understanding of the neuronal mechanisms underlying anxiety expression, this study could provide a biomarker of anxiety with diagnostic and therapeutic implications.

ELIGIBILITY:
Inclusion Criteria:

* Social anxiety disorder as defined in DSM-5
* Full understanding of the protocol
* Obtaining informed consent from study subjects before or at inclusion at the latest
* Being registered in the french national health insurance service (Sécurité Sociale) (or equivalent)

Exclusion Criteria:

* Active medical co-morbidity including severe hypertension, cardiac insufficiency, Raynaud syndrome, diabetes mellitus, renal insufficiency, adrenal insufficiency, Cushing syndrome and epilepsy
* Severe neurological co-morbidity, including but not limited to Parkinson's disease and multiple sclerosis
* Long-term corticotherapy
* History of significant head injury, defined by loss of consciousness
* Being diagnosed with another major psychiatric condition (DSM5) including bipolar disorder and schizophrenia or substance/alcohol use disorder; with the exception of major depressive disorder and nicotine use disorder
* Suicidal risk evaluated as moderate to high in the MINI questionnaire
* initiation of a psychotropic treatment or change in the dose of ongoing psychotropic treatment within 3 days prior to each visit and including:

  1. antidepressant treatments with selective serotonin recapture inhibitors, serotonin and norepinephrine inhibitors, alpha2-presynaptic adrenoreceptors (mirtazapine, mianserin), tricyclic
  2. anxiolytic drugs including benzodiazepines and anti-histamine
  3. antipsychotic drugs
* Acute alcohol intake 2 days prior to each visit (inclusion, experimental sessions)
* Pregnancy or breastfeeding.
* Ongoing hospitalization without consent (decision of a third-party: medical, justice)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
Change in power of slow oscillations in prefrontal EEG recordings during anticipation relative to baseline | During the 5 minutes before oral presentation and during the 1 hour rest period
  The change in power of PFC 2-6 Hz oscillations between the 5-minutes waiting period before oral presentation and the recovery period will be computed as a ratio.
  Detection of exaggerated 2-6Hz oscillations in prefrontal cortex during anxious anticipation is the primary aim of this study.

SECONDARY OUTCOMES:
Duration of prefrontal slow oscillations epochs during anticipation | During the 5 minutes before oral presentation
  Time-frequency analysis will be performed to determine the duration of 2-6Hz prefrontal oscillations epochs and total duration of these oscillations within experimental period. Significant oscillatory epochs will be defined using power ratios. These metrics will be used in order to assess the neurobiological and clinical relevance of this biomarker.

OTHER OUTCOMES:
Change in power of slow oscillations in prefrontal EEG recordings during presentation relative to baseline | During the 5 minutes oral presentation and during the 1 hour rest period.
  The change in power of PFC 2-6 Hz oscillations between the 5-minutes oral presentation and the recovery period will be computed as a ratio.
Duration of prefrontal slow oscillations epochs during presentation | During the 5 minutes oral presentation
  Time-frequency analysis will be performed to determine the duration of 2-6Hz prefrontal oscillations epochs and total duration of these oscillations within experimental period. Significant oscillatory epochs will be defined using power ratios.
Correlation between prefrontal slow oscillations power during anticipation and anxiety score | During the 5 minutes before oral presentation
  Correlation will be calculated between PFC 2-6 Hz oscillations power and the visual Analogue anxiety score during the 5 minutes period before presentation.
Correlation between prefrontal slow oscillations power during presentation and anxiety score | During the 5 minutes oral presentation
  Correlation will be calculated between PFC 2-6 Hz oscillations power and the visual Analogue anxiety score during presentation.
Correlation between prefrontal slow oscillations duration during anticipation and anxiety score | During the 5 minutes before oral presentation
  Correlation will be calculated between PFC 2-6 Hz oscillations duration and the visual Analogue anxiety score during the 5 minutes period before presentation.
Correlation between prefrontal slow oscillations duration during presentation and anxiety score | During the 5 minutes oral presentation
  Correlation will be calculated between PFC 2-6 Hz oscillations duration and the visual Analogue anxiety score during presentation.
Correlation between prefrontal slow oscillations power during anticipation and trait anxiety | During the 5 minutes before oral presentations (PFC oscillations power) and prior to inclusion (STAI-B rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during the 5 minutes before presentation and STAI-B scores
Correlation between prefrontal slow oscillations power during presentation and trait anxiety | During the 5 minutes oral presentation (PFC oscillations power) and prior to inclusion (STAI-B rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during presentation and STAI-B scores
Correlation between prefrontal slow oscillations duration during anticipation and trait anxiety | During the 5 minutes before oral presentation (PFC oscillations duration) and prior to inclusion (STAI-B rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during the 5 minutes before presentation and STAI-B scores
Correlation between prefrontal slow oscillations duration during presentation and trait anxiety | During the 5 minutes oral presentation (PFC oscillations duration) and prior to inclusion (STAI-B rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during presentation and STAI-B scores
Correlation between prefrontal slow oscillations power during anticipation and state anxiety | During the 5 minutes before oral presentation (PFC oscillations power) and prior to inclusion (STAI-A rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during the 5 minutes before presentation and STAI-A scores
Correlation between prefrontal slow oscillations power during presentation and state anxiety | During the 5 minutes oral presentation (PFC oscillations power) and prior to inclusion (STAI-A rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during presentation and STAI-A scores
Correlation between prefrontal slow oscillations duration during anticipation and state anxiety | During the 5 minutes before oral presentation (PFC oscillations duration) and prior to inclusion (STAI-A rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during the 5 minutes before presentation and STAI-A scores
Correlation between prefrontal slow oscillations duration during presentation and state anxiety | During the 5 minutes oral presentation (PFC oscillations duration) and prior to inclusion (STAI-A rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during presentation and STAI-A scores
Correlation between prefrontal slow oscillations power during anticipation and levels of social anxiety | During the 5 minutes before oral presentation (PFC oscillations power) and prior to inclusion (LSAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during the 5 minutes before presentation and LSAS scores
Correlation between prefrontal slow oscillations power during presentation and levels of social anxiety | During the 5 minutes oral presentation (PFC oscillations power) and prior to inclusion (LSAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during presentation and LSAS scores
Correlation between prefrontal slow oscillations duration during anticipation and levels of social anxiety | During the 5 minutes before oral presentation (PFC oscillations duration) and prior to inclusion (LSAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during the 5 minutes before presentation and LSAS scores
Correlation between prefrontal slow oscillations duration during presentation and levels of social anxiety | During the 5 minutes oral presentation (PFC oscillations duration) and prior to inclusion (LSAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during presentation and LSAS scores
Correlation between prefrontal slow oscillations power during anticipation and levels of general anxiety | During the 5 minutes before oral presentation (PFC oscillations power) and prior to inclusion (BAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during the 5 minutes before presentation and BAS scores
Correlation between prefrontal slow oscillations power during presentation and levels of general anxiety | During the 5 minutes oral presentation (PFC oscillations power) and prior to inclusion (BAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during presentation and BAS scores
Correlation between prefrontal slow oscillations duration during anticipation and levels of general anxiety | During the 5 minutes before oral presentation (PFC oscillations duration) and prior to inclusion (BAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during the 5 minutes before presentation and BAS scores
Correlation between prefrontal slow oscillations duration during presentation and levels of general anxiety | During the 5 minutes oral presentation (PFC oscillations duration) and prior to inclusion (BAS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during presentation and BAS scores
Correlation between prefrontal slow oscillations power during anticipation and depression levels | During the 5 minutes before oral presentation (PFC oscillations power) and prior to inclusion (MARDS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during the 5 minutes before presentation and MADRS scores
Correlation between prefrontal slow oscillations power during presentation and depression levels | During the 5 minutes oral presentation (PFC oscillations power) and prior to inclusion (MARDS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations power during presentations and MADRS scores
Correlation between prefrontal slow oscillations duration during anticipation and depression levels | During the 5 minutes before oral presentation (PFC oscillations duration) and prior to inclusion (MARDS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during the 5 minutes before presentation and MADRS scores
Correlation between prefrontal slow oscillations duration during presentation and depression levels | During the 5 minutes oral presentations (PFC oscillations duration) and prior to inclusion (MARDS rating)
  Correlation will be calculated between PFC 2-6 Hz oscillations duration during presentation and MADRS scores

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Doumy, MD, Principal Investigator — Centre Hospitalier Charles Perrens, Bordeaux; INRA NutriNeuro, Bordeaux; Université de Bordeaux, France; Alexandra Bouvard, MD, Principal Investigator — Centre Hospitalier Charles Perrens, Bordeaux; Université de Bordeaux, France; Cyril Herry, PhD, Study Director — Neurocentre Magendie, Inserm U1215, Bordeaux, France; Cyril Dejean, PhD, Principal Investigator — Neurocentre Magendie, Inserm U1215, Bordeaux, France; Thomas Bienvenu, PhD, Principal Investigator — Centre Hospitalier Charles Perrens, Bordeaux; Neurocentre Magendie, Inserm U1215, Bordeaux, France; Jacques Taillard, MS, Principal Investigator — GENPHASS, CHU de Bordeaux; Bruno Aouizerate, MD-PhD, Study Chair — Centre Hospitalier Charles Perrens, Bordeaux; INRA NutriNeuro, Bordeaux; Université de Bordeaux, France
Locations (1):
- GENPHASS, SANPSY, CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No